CLINICAL TRIAL: NCT01251263
Title: Prevention of Menstrual Migraines: Effects of Estrogen Add-back During the HFI in Patients Using Continuous Oral Contraceptives.
Acronym: Estradiol/MAM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scott and White Hospital & Clinic (Other)
Responsible Party: Patricia Sulak, MD/Principal Investigator, Scott and White Hospital & Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 90304
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-10

CONDITIONS: Menstrual Migraines; Menstrual Bleeding; Menstrual Spotting
Keywords: headaches; migraines; breakthrough bleeding; breakthrough spotting; menstrually associated migraines; breakthrough bleeding or breakthrough spotting
MeSH Terms: conditions — Metrorrhagia; Headache; Migraine Disorders | interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Other): Cyclic OC users prior to initiating study OC. Estradiol or placebo given in a certain sequence depending on the randomization.
  Interventions: Drug: Estradiol or Placebo
- Group 2 (Other): Spontaneous ovulation group prior to initiating study OC. Estradiol or placebo given in a certain sequence depending on the randomization.
  Interventions: Drug: Estradiol or Placebo

INTERVENTIONS:
Drug: Estradiol or Placebo — Estradiol 1mg twice daily or placebo starting on the last day of OC and continuing during the HFI (total of 9 doses).
  Arms: Group 1
Drug: Estradiol or Placebo — Estradiol 1mg will be taken twice daily starting with the last day of pills and the 4 days of the HFI(total of 9 doses)
  Arms: Group 2

SUMMARY:
This study will examine the combined effects of a continuous oral contraceptive (OC) regimen with supplemental estradiol therapy on headache severity and occurrence in subjects with documented Menstrually Associated Migraines (MAMs). The subjects enrolling in the study will have cyclic menses either due to spontaneous ovulation or use of cyclic hormonal contraception (pill, patch, or ring). Enrolled subjects will start a continuous OC regimen following two baseline menstrual cycles. If breakthrough bleeding/spotting (BTB/BTS) occurs, the subject will institute a 4-day hormone-free interval (HFI). In an attempt to prevent/lessen the severity of headache during the HFI, subjects will be randomized to oral estradiol or placebo during this period. If no BTB/BTS occurs after 80 days of continuous pills, the subject will institute a 4-day HFI during which they will be randomized into estradiol or placebo groups.

The purpose of this research study is to examine the effects of continuous oral contraceptive pills and oral estradiol on headaches that occur around the time of your period. Many woman take continuous oral contraceptive pills (OC) and when OCs are stopped they may get headaches. This study will examine if taking estradiol around the time of the period will affect the headache, and how it will be affected.

This study is a prospective trial. A subject's participation will last approximately 32 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women may be on birth control pill (OC), patch or vaginal ring taken in the traditional 21/7 or 24/4 manner, which means that every month they have a period. If they are taking it continuously (without a period), you must be willing to take your birth control 21/7 for 2 months.
* If you are not on OC's, patch or vaginal ring you must have a period every 21-40 days.
* You must not want to get pregnant for 12 months.
* Women who have headaches around the time of their period.

Exclusion Criteria:

* BMI >38
* If you smoke and are age 35 years old or greater or if you are under 35 years old and smoke over 10 cigarettes a day.
* If you have or had an aura with your headaches. (An aura is a temporary sensation, like bright lights that come before you experience the headache)
* Headaches are not occuring during the time of your period.
* Blood Pressure > 140/90 or you take more than a single antihypertensive medication (excluding diuretics) and are age 40 or greater.
* Contraindications to combination estrogen/progestin hormonal contraceptives.
* Desire to become pregnant in the next 12 months.
* Stroke
* Breast Cancer
* Blood clots in your legs, lung or anywhere else in your body.
* Diabetes Mellitus
* Heart Attack
* Liver Disease
* Systemic Lupus Erythematosus

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | 32 weeks
  Comparing baseline menstrually associated migraines(MAMs) to headache occurance and severity after the implementation of continuous OC therapy.

SECONDARY OUTCOMES:
Secondary Outcome Measure | 32 weeks
  Compare effect of estradiol versus placebo on MAMs severity and duration.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia J Sulak, MD, Principal Investigator — Scott and White Healthcare
Locations (1):
- Scott and White Hospital & Clinic, Temple, Texas, United States